CLINICAL TRIAL: NCT04552886
Title: A Phase I Study of Th-1 Dendritic Cell Immunotherapy in Combination With Standard Chemoradiation for the Adjuvant Treatment of Adult Glioblastoma
Brief Title: Dendritic Cell Vaccination With Standard Postoperative Chemoradiation for the Treatment of Adult Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Cooper Health System (Other)
Collaborators: Baylor College of Medicine (Other); Philadelphia College of Osteopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8148
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: The study will be constructed in a 3+3 algorithm for three steps of dose escalation for a novel GBM-targeting dendritic cell vaccine with rigorous and mandatory safety monitoring.
Masking Description: Patients, clinicians, investigators and support staff will be aware of the enrollment status of patients in this phase I trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dendritic cell vaccine: Starting dose (Experimental): This arm will evaluate the safety of administering a total dendritic cell dose of 3.5 x 10^6. A total of 3-6 patients will be enrolled with this dose. If this dose is associated with unacceptable side effects, as detailed in the study protocol, no further patients will be enrolled at this dose.
  Interventions: Biological: TH-1 Dendritic Cell Immunotherapy
- Dendritic cell vaccine dose de-escalation (Experimental): If unacceptable side effects, as detailed in the study protocol, are identified at a total dose of 3.5 x 10^6, then a cohort of 3-6 enrolled patients will receive a de-escalated total dendritic cell dose of 1.75 X 10^6.
  Interventions: Biological: TH-1 Dendritic Cell Immunotherapy
- Dendritic cell vaccine dose escalation one (Experimental): If no unacceptable side effects, as detailed in the study protocol, are identified at a total dose of 3.5 x 10^6, then a cohort of 3-6 enrolled patients will receive an escalated total dendritic cell dose of 7.0 X 10^6.
  Interventions: Biological: TH-1 Dendritic Cell Immunotherapy
- Dendritic cell vaccine dose escalation two (Experimental): If no unacceptable side effects, as detailed in the study protocol, are identified at a total dose of 7.0 x 10^6, then a cohort of 3-6 enrolled patients will receive an escalated total dendritic cell dose of 1.4 X 10^7.
  Interventions: Biological: TH-1 Dendritic Cell Immunotherapy

INTERVENTIONS:
Biological: TH-1 Dendritic Cell Immunotherapy — Adult patients with histopathologically diagnosed glioblastoma will be eligible for this novel, personalized dendritic cell vaccine after completing standard of care chemoradiation.

SUMMARY:
Effective treatments are desperately needed for glioblastoma (GBM) patients. This phase I clinical trial assesses the safety of a novel personalized dendritic-cell vaccine administered to GBM patients shortly after completing standard-of-care treatments. Secondary outcomes will evaluate patient progression-free survival and overall survival.

DETAILED DESCRIPTION:
This is a single arm (non-randomized) first-in-man pilot study to evaluate the safety and feasibility of delivering a dendritic cell vaccine in nine to twenty-four (n=9-24) adult patients diagnosed with glioblastoma (GBM) after undergoing neurosurgical tumor resection, and in whom a neuropathological diagnosis has been established. Standard of care chemotherapy and radiation therapy shall be followed as per routine neuro-oncologic paradigms after which patients enrolled into this study will receive a personalized vaccine beyond standard of care. Effective adjuvant therapies are urgently needed for these patients given that standard of care is rarely successful in preventing recurrence among GBM patients, nor death among relapsed patients with this very poor-prognosis tumor type. The study is constructed in a 3+3 algorithm for three steps of dose escalation with rigorous and mandatory safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 years and older
4. Diagnosed with glioblastoma (GBM) deemed to be potentially resectable and who are deemed to be good candidate for postoperative adjuvant chemo and radiation therapy. This may include patients whose tumors are deemed suitable for gross total resection as well as patients whose tumors are deemed partially resectable and who undergo partial resection followed by adjuvant therapy. [neoadjuvant therapy is rarely if ever given]..
5. Ability to adhere to the bi-weekly injections of DC vaccine regimen
6. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 12 weeks following discontinuations of last vaccination. Must have a negative serum pregnancy test prior to first treatment.
7. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner during study participation and for an additional 12 weeks following discontinuations of last vaccination.
8. Presented at Tumor Board for review and consensus of Multidisciplinary group to proceed with enrollment.
9. Adequate kidney, liver, bone marrow function, and immune function, as follows:

   1. Hemoglobin ≥ 8.0 gm/dL
   2. Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
   3. Platelet count ≥ 100,000 /mm3
   4. Lymphocyte count greater than 500/L
   5. Glomerular filtration rate (GFR) > 60 mL/min/m2 and Creatinine < 1.5mg/dl

   i. For males = (140 - age[years]) x (body weight [kg]) (72) x (serum creatinine [mg/dL] ii. For females = 0.85 x male value f. Total bilirubin ≤ 1.5 times upper limit of normal (ULN), g. Aspartate transaminase AST (SGOT) and alanine aminotransferase ALT (SGPT) ≤ 2.5 times the ULN h. Albumin >2g/dL i. (IgM), surface antibody and antigen, Hepatitis B and C antibody. j. Negative HIV status
10. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.

Exclusion Criteria:

1. Locally advanced tumors deemed unresectable and/or recurrent tumors after prior vaccination.
2. Use of non-standard post-operative treatment regimen, as defined by the Stupp protocol: postoperative chemoradiation and initiation of temozolomide (TMZ). The use of a tumor treatment field (TTF) device with adjuvant TMZ is at the discretion of the investigator.
3. Female patients who are pregnant, breast feeding, or of childbearing potential without a negative pregnancy test prior to baseline. Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
4. Patients unwilling or unable to comply with the protocol or provide informed consent.
5. Any severe or uncontrolled medical condition or other condition that could affect participation in this study, including but not limited to: hyper/hypothyroidism, systemic autoimmune disorders, untreated viral hepatitis or autoimmune hepatitis.
6. Concurrent or expected need for therapy with corticosteroids during the vaccination phase of the study.
7. Treatment with another investigational drug or other intervention outside of the prespecified standard of care for GBM.
8. Patients suffering from active HIV disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Safety and potential toxicity of Th-1 dendritic cell immunotherapy | Two years
  Patients will be monitored for adverse events as dictated by CTCAE version 5.

SECONDARY OUTCOMES:
Overall survival of patients receiving Th-1 dendritic cell immunotherapy | Minimum 2 years from time of diagnosis
  Length of survival for patients who receive this vaccine will be tabulated.
Progression-free survival of patients receiving Th-1 dendritic cell immunotherapy | Minimum 2 years from time of diagnosis
  If there is tumor recurrence, the time from diagnosis until recurrence will be collected

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cooper University Hospital, Camden, New Jersey
  - Memorial Hermann- Texas Medical Center, Houston, Texas